CLINICAL TRIAL: NCT03411057
Title: Mindfulness Based Stress Reduction in Rheumatic Diseases
Acronym: MBSR
Status: Terminated | Type: Observational
Why Stopped: PI is leaving the institution
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00147638
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Scleroderma
Keywords: Mindfulness; Mindfulness Based Stress Reduction; Rheumatoid Arthritis; Anxiety; Depression; Psoriatic Arthritis; scleroderma
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Scleroderma, Diffuse; Anxiety Disorders; Depression | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum will be collected at research visits within one-month the Mindfulness Based Stress Reduction (MBSR) course start and end. Serum will be used to analyze levels of C-Reactive Protein (CRP) and pro-inflammatory cytokines (Mesoscale 4-plex pro-inflammatory panel 1).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mindfulness Based Stress Reduction (MBSR): Inflammatory Arthritis (Rheumatoid Arthritis, Psoriatic Arthritis) and scleroderma participants in this group will attend an 8 week MBSR course. The MBSR course meets once per week for 2.5 hours with a 4-hour retreat on week 8.
  Interventions: Behavioral: Mindfulness Based Stress Reduction (MBSR)
- Control: Rheumatoid Arthritis, Psoriatic Arthritis, and scleroderma participants in this group will watch an educational stress reduction video (10 minutes).
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction (MBSR) — An interactive form of meditation that includes gentle yoga.
  Groups: Mindfulness Based Stress Reduction (MBSR)
Other: Control — Standard of care including an educational video.
  Groups: Control

SUMMARY:
This study will assess the mental health and clinical benefits of Mindfulness Based Stress Reduction (MBSR) in patients with rheumatic disease who have anxiety or depression. MBSR, an interactive form of meditation that includes gentle yoga, will be taught by a certified instructor over an eight-week period. Mental health surveys will be conducted within one month of the study start and end as well as mid-course. Clinical assessments will be conducted within one-month of the study start and end.

DETAILED DESCRIPTION:
Participation in the study entails completing a baseline and 1-month post MBSR follow up research appointment. A baseline research appointment must occur within 30 days (+/- 15 days) of the MBSR start. The 1 month follow up appointment must be completed within 30 days (+/- 15 days) after the MBSR course end. At each research appointment, disease activity, patient reported outcome measures (PROMs), and blood will be collected for future analysis. Patients will also be asked to complete the PROMs through an online survey platform using email, at MBSR course start, week 4 of the MBSR course, and at MBSR course end. Participants in the MBSR arm will also be recommended to perform self-directed meditation for 20-40 minutes per day, on off-days, throughout the 8-week session, as is typical for the MBSR course. Compliance with home meditation will be recorded on a take-home "practice" sheet that will be collected each week during the MBSR course.

If patients do not wish to participate in the MBSR course but are willing to participate in the study as a control, patients may also be consented. Controls will be asked to attend a baseline and 3-month research appointment where disease activity, PROMs, and blood donation would be obtained. Participants will also be asked to fill out PROMs (online) at 4 weeks. If a patient does not wish to participate in either arm of the MBSR study, patient will continue with routine psychological care for patient's anxiety and depression.

Blood samples will be collected at the baseline research appointment and the follow up research appointment, if the patient is willing. These samples will be drawn and banked for future analysis of inflammatory markers and cytokine expression.

Participants will be sent a health care usage survey after 3 months (coinciding with research visit 2; 1 month post-MBSR research visit or 3-month follow up research visit if control). Health care usage will continue to be screened for up to 1 year post research visit 1 via the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* Established patients in the Johns Hopkins Bayview Rheumatology clinic
* Rheumatoid Arthritis per the American College of Rheumatology (ACR) and European League Against Rheumatism (EULAR) 2010 classification criteria
* Psoriatic Arthritis per the Classification Criteria for Psoriatic Arthritis (CASPAR) or physician-diagnosis
* Scleroderma per the ACR/EULAR 2013 classification criteria or physician-diagnosis
* New onset of Comorbid anxiety and/or depression
* Participants must speak English
* Participants must be able to attend a weekly (8 weeks total) Mindfulness Based Stress Reduction course as well as routine follow up appointments in the rheumatology clinic
* Participants must have insurance

Exclusion Criteria:

* Patients who routinely perform mindfulness based practices and any other form of meditation, including moving meditations such as yoga
* Patients who are not physically able to sit through weekly sessions that are 2.5 hours in length or a final meditative retreat of 4-hours duration
* Patients with alcohol or substance use disorders within the past 6 months
* Current, or previous history of psychotic disorders or bipolar disorder
* Patients who are actively suicidal
* Patients on greater than 10 mg of prednisone daily on a chronic basis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Established patients of the Johns Hopkins Arthritis and Scleroderma Centers
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
Change in anxiety | Baseline, midcourse (approximately 4 weeks), post course (approximately 8-12 weeks)
  Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety Scale (8a). The PROMIS Anxiety Scale is measured as a t score with a t-score range from 41 (less anxious) to 80 (highly anxious). For most PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10.
Change in Self-Efficacy (Symptoms) | Baseline, midcourse (approximately 4 weeks), post course (approximately 8-12 weeks)
  Patient Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy Scale 8a. The PROMIS Self-Efficacy (Symptoms) Scale is measured as a t score with a t-score range from 41 (less efficacious) to 80 (highly efficacious). For most PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10.
Change in Self-Efficacy (Emotions) | Baseline, midcourse (approximately 4 weeks), post course (approximately 8-12 weeks)
  Patient Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy Scale 8a. The PROMIS Self-Efficacy (Symptoms) Scale is measured as a t score with a t-score range from 41 (less efficacious) to 80 (highly efficacious). For most PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10.

SECONDARY OUTCOMES:
Change in Clinical Disease Activity Index (CDAI) | Baseline and post course (approximately 8-12 weeks)
  The CDAI is calculated by the formula, CDAI = swollen joint count (28 sites) + tender joint count (28 sites) + patient global assessment (0-10; 10= severe) + evaluator global assessment (0-10; 10=severe). The total range is 0 to 76. Higher scores indicate more severe disease activity. Remission is considered less than 2.8, mild disease 2.8 to 10, moderate disease 10 to 22, and severe disease greater than 22.
Change in C-Reactive Protein (CRP) | Baseline and post course (approximately 8-12 weeks)
  A value of 0-0.5 mg/dL indicates a normal range. Values greater 0.5 mg/dL indicate elevated degrees of inflammation.
Change in Medsger Disease Severity Score (Composite Measure of Scleroderma Disease Activity) | Baseline and post course (approximately 8-12 weeks)
  The Medsger Severity Score is a composite measure for scleroderma disease activity comprised of the following sub-domains: general, peripheral vascular, skin, join/tendon, muscle, GI tract, lung, heart, kidney. Each sub-domain ranges from 0-4 (4=worse). The total Medsger Disease Severity Score is a sum of the subdomains and ranges from 0-36 (36= worse).

CONTACTS AND LOCATIONS:
Overall Officials: Dana DiRenzo, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Asthma and Allergy Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No